CLINICAL TRIAL: NCT04605341
Title: Comparative Study Between Miniplate and Buried k Wires in Management of Metacarpal Fractures
Brief Title: Miniplate Versus k Wires in Management of Metacarpal Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mina kamal, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: miniplate,k wires and union
Record Dates: First submitted 2020-09-12; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-09

CONDITIONS: Metacarpal Fracture
MeSH Terms: interventions — Bone Wires

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group one (Active Comparator): patient with metacarpal fracture that will use minipate for fixation
  Interventions: Device: miniplate
- gruop two (Active Comparator): patient with metacarpal fracture that will use buried k wires for fixation
  Interventions: Device: miniplate

INTERVENTIONS:
Device: miniplate — comparison between k wires and miniplate in metacarpal fractures
  Other Names: k wires

SUMMARY:
To compare between buried k wires and miniplate in management of metacarpal fracture.

DETAILED DESCRIPTION:
Fractures of the carpals, metacarpals and phalanges account for approximately 15-19% of fractures in adults, with 59% of these occurring in the phalanges, 33% in the metacarpals and 8% in the carpal bones [1]. The single most common fracture site in the hand is the sub capital region of the fifth metacarpal bone (boxer's fracture) [2], which usually results from a direct blow to the metacarpal head [3]. Most hand fractures are caused by accidental falls or other sports-related injuries [4]. Hand fractures are among the most common fractures of upper extremity [5, 6]. Hand fractures can be treated conservatively or surgically, depending on the severity, location and type of fracture. The main objective of both operative and non-operative treatments is to provide fracture stability for early mobilization [7]. Surgical fixation is mainly indicated for displaced fractures because casts are often not sufficient to maintain reduction [8]. Open reduction with internal fixation (ORIF), using pins or plates, has historically been used to stabilize hand fractures which have rotational deformity or lateral angulation [9]. Open reduction may result in scarring, joint stiffness and tendon adhesion [7]. Closed reduction with internal fixation (CRIF), using percutaneous K wire or screws, is now used to treat the majority of unstable closed simple hand fractures [10]. It is generally considered percutaneous Kirschner wire (K wire) fixation may not provide adequate stabilization to allow for early mobilization [8] .

ELIGIBILITY:
Inclusion Criteria:

1. Age: ( 20-60) years,
2. Fresh (fixed within 3 days),
3. Single or multiple fractures of metacarpals.

Exclusion Criteria:

1. Pathological fracture,
2. Major systemic illness, malignancy,
3. Patient on drugs affecting fracture healing like steroid, anticancer drugs,
4. Polytrauma patients,
5. Extensive comminution of the metacarpal or phalanx detected pre- or intra-operatively,
6. Dislocations at either end of the fractured bone
7. Parents/guardians/patients not willing to participate in study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
miniplate,buried k wires and union | 6 month
  • To compare between union and healing in metacarpal fracture fixation by miniplate versus buried intramedullary k. wires by imaging using anteroposterior and lateral and oblique views x ray to determine union and healing by seeing bridging callus in two or more cortices

SECONDARY OUTCOMES:
Range of motion | 6 month
  • Range of motion using Functional range of motion (FROM) is defined as the minimum ROM necessary to comfortably and effectively perform ADL.